CLINICAL TRIAL: NCT02500966
Title: A Randomized Study to Evaluate the Safety, Efficacy and Quality of Life of a New Device to Prevent Cervical Stenosis After LEEP in High Grade Cervical Dysplasia
Brief Title: How to Avoid Cervical Stenosis After LEEP in High Grade Cervical Dysplasia?
Acronym: DUDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BarretosCH - DUDA
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2018-06

CONDITIONS: Stenosis Cervix
Keywords: Cervical Intraepithelial Neoplasia; stenosis; cervix; medical device; inventories; Uterine Cervix; Intrauterine Devices; intrauterine; conization; loop electrosurgical excision
MeSH Terms: conditions — Uterine Cervical Dysplasia; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DUDA device (Experimental): The number of patients to be recruited in this arm will be 145. Note: The first twenty-five patients who will be included in the study will be allocated in the intervention arm to safety analysis (phase 1); after that all eligible candidates will be randomized 1:1 (phase 2).
  Procedure: Loop Electrosurgical Excision Procedure (LEEP) followed by implantation of the device called DUDA (plastic device developed in barretos cancer hospital that will be placed after conization. It has 2.5 cm in length and 5mm in diameter and remains within the endocervical canal for 30 days and is set at 4 points with nonabsorbable sutures in the ectocervix.)
  Interventions: Device: DUDA device; Procedure: LEEP
- Control group (Active Comparator): The number of patients to be recruited in this arm will be 120.
  Procedure: Loop Electrosurgical Excision Procedure (LEEP) without DUDA device
  Interventions: Procedure: LEEP

INTERVENTIONS:
Device: DUDA device — Insertion DUDA device
  Arms: DUDA device
Procedure: LEEP — Loop Electrosurgical Excision Procedure

SUMMARY:
Cervical stenosis may occur in up to 19% after conization. It is a cause of infertility and amenorrhea. This study will test a new device named DUDA Device ("Dispositivo Uterino para dilatar canal endocervical") placed just after the conization, in order to evaluate the safety, efficacy and quality of life.

DETAILED DESCRIPTION:
This device has the potential to improve outcomes by means of a significant stenosis reduction and maintain patency of the endocervical canal to view the squamo-columnar junction (SCJ) of the cervix during follow-up of this patient.

ELIGIBILITY:
Inclusion Criteria:

* High Grade Cervical Dysplasia, Grades 2 and 3, in the biopsy cervical
* Patient eligible for conization
* Patient must consent for the appropriate surgery
* Patient must have Gynecologic Oncology Group (GOG) performance status of 0, 1
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Pregnancy
* Previous conization
* limited comprehension of the study
* the risk of the American Society of Anesthesiologists, III or IV
* HIV or immunodepression
* Patients with a history of the invasive malignancies

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2015-08; Primary Completion 2018-06 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Safety (two adverse events Grade 3 or 4 (CTCAE v. 4.0) or a single adverse event Grade 5) | 3 months
  The main safety events to be considered in this analysis are vaginal bleeding and uterine infection. The device is considered unsafe and consequently disrupted the study if a two adverse events Grade 3 or 4 (CTCAE v. 4.0) or a single adverse event Grade 5 related to the procedure/device happens during the phase 1.
Cervical stenosis | 6 months
  Stenosis of the endocervical canal (early and late) will be assessed by clinical information and physical examination at each visit to the hospital after surgery. The participant will be asked about the menstrual flow and dysmenorrhea during history taking. On physical examination, after the visualization of the cervix through the speculum examination, the doctor will check the channel permeability introducing a hysterometer through it. The difficulty of introducing the hysterometer 2.5mm the channel will be scored according to the following scale:
  Possible passage of hysterometer? () No difficulty () Little difficult, however possible passage of hysterometer () Unable to pass

SECONDARY OUTCOMES:
Pain Scales | 6 months
  The quality of life will be evaluated through questionnaires by the Functional Assessment of Cancer Therapy - Cervix Cancer (FACT-Cx) and the universal pain assessment tools that include international scale and pain visual analogue (EVA), numerical visual pain scale (EVN) and faces pain scales (EF).
Complications | 30 days
  It will be evaluated during the following returns and described as any event related directly to the use of DUDA device as metrorrhagia and uterine infection.
View of the squamo-columnar junction (SCJ) of the cervix | 6 months
  It will be assessed during the examination of colposcopy

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Reis, PHD, Study Director — Director of the Teaching and Research Institute - Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil